CLINICAL TRIAL: NCT03049631
Title: The Reciprocal Interactions Between Red Raspberry Polyphenols and Gut Microbiome Composition Affect Insulin Sensitivity
Brief Title: Red Raspberry Polyphenols on Gut Microbiome
Acronym: RRB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB2016-136
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subjects; Pre-diabetes
Keywords: Pre-diabetes; red raspberry; fructooligosaccharide; metagenomics; polyphenol bioavailability; glycemic response; insulin response
MeSH Terms: conditions — Glucose Intolerance | interventions — fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raspberry and fructooligosaccharide (Active Comparator): Red raspberries (1 cup equivalent) with fructooligosaccharide (8 g)
  Interventions: Dietary Supplement: Raspberry and fructooligosaccharide
- Raspberry (Experimental): Red raspberries (1 cup equivalent)
  Interventions: Dietary Supplement: Raspberry

INTERVENTIONS:
Dietary Supplement: Raspberry and fructooligosaccharide — Red raspberries (1 cup equivalent) with fructooligosaccharide (8 g)
  Arms: Raspberry and fructooligosaccharide
Dietary Supplement: Raspberry — Red raspberries (1 cup equivalent)
  Arms: Raspberry

SUMMARY:
The primary objective aims are to assess the effects of regular consumption of red raspberries (RRB) with and without fructooligosaccharide (FOS) on the composition of the gut microbiota after 4 week intake and in parallel characterize plasma and urine metabolite profiles examining qualitative and quantitative intervention associated changes.

DETAILED DESCRIPTION:
The study will be performed as a single-blinded, randomized, crossover manner. Thirty subjects (20 insulin resistant subjects and 10 healthy subjects) will be randomly assigned into one of two sequences: sequence A (n=15) will be RRB then RRB+FOS (which means subject will consume only RRB (125 g/day(d) (equivalent to 1 cup fresh RRB)) with breakfast for 4 weeks, and then after a 4-week washout period, that subject will consume the RRB with FOS (125 g/d RRB and 8 g/d FOS) for 4 weeks); sequence B (n=15) will be RRB+FOS then RRB (which means subject will receive the RRB with FOS for 4 weeks, a 4-week washout, and then the RRB for another 4-week). At the beginning and end of each 4-week treatment, subjects will undergo a 6-h Study Day (4 study days in 12-week study duration) followed by a 1-h next morning follow-up visit.

Subjects will be required to meet several inclusion and exclusion criteria, which will be assessed through online survey and on-site clinic assessments, including questionnaires, blood analysis and anthropometric measures. Eligible subjects will be invited to participate in the study. Each subject will be asked to come for 1 Screening Visit, 4 dinner pick-ups (the day before each Study Day), 4 Study Days and 6 Weekly Meetings.

During the Screening Visit, subjects will read, sign and date a written Institutional Review Board approved Informed Consent Form prior to performing any study procedure. And then they will be assessed their qualification, instructed on the process for completing study questionnaires and counseled to restrict intake of colored plant foods rich in phytonutrients the 3 days prior to each Study Day. They will be asked to restrict alcohol intake, coffee/tea/ caffeinated beverage intake and moderate / vigorous physical activity and to drink plenty of water to maintain hydration in the 24 h prior to each Study Day. They will be instructed to come to the Clinical Nutrition Research Center (CNRC) the day before each Study Day to pick up their dinner meal and evening snack. Subjects will be asked to get at least 7 hours sleep and to come to the CNRC after a 10-h overnight fasting on each Study Day.

Each Study Day will require subjects to be in the clinic for ~7 h to complete all baseline and post challenge beverage testing procedures, including a 6 h study day and a 1 h next morning follow-up visit. Subjects will be evaluated for compliance with the protocol (diet, exercise, sleep, fasting), have their body weight and blood pressure measured, ingest a cup of red raspberry drink (250 g RRB (equivalent to 2 cups fresh RRB) and 64 g glucose) and their blood, urine and feces samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking1 man or woman, 20-60 years of age, inclusive
2. Group 1 must have a fasting blood glucose between 100-125 mg/dL and inulin ≥ 8 μIU/mL
3. Group 2 will have a fasting blood glucose below 100 mg/dL and the homeostasis model assessment method of insulin resistance (HOMA-IR) [glucose (μmol/L) × insulin (μunits/μL)/22.5] value less than 1
4. Judged to be in good health on the basis of the medical history
5. Able to provide informed consent and comply with study procedures
6. Able to comply to the study instructions (including dietary restrictions, consumption of study beverage, records of food diary and GI-tract questionnaire, sample collection procedure and study visit schedule)
7. Able to maintain your usual physical activity pattern
8. Able to abstain from alcohol consumption and avoid vigorous physical activity for 24 hours prior to and during study visit

Exclusion Criteria:

1. Systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg at screening visit.
2. Major trauma or a surgical event within 2 months or longer depending on trauma or event and after consultation with PI.
3. Weight change ≥4.5 kg (9.9 lbs) within 2 months
4. Presence of chronic constipation, diarrhea or other chronic gastrointestinal complaint (e.g. irritable bowel syndrome)
5. Had gastrointestinal barium opaque meal within 3 months
6. History or presence of clinically important endocrine, cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, or biliary that, in the opinion of the investigator, could interfere with the interpretation of the study results
7. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer
8. History of extreme dietary habits, as judged by the investigator (e.g., Atkins diet, etc.)
9. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
10. Vegan or other extreme dietary regimens as judged by the investigator.
11. Has a known intolerance or sensitivity to any ingredients in the study products
12. Has used antibiotics within the previous 2 months
13. Has used prebiotics, probiotics, or drugs active on gastrointestinal motility, or a laxative of any class within 1 month
14. Has used medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, hypoglycemic medications, and systemic corticosteroids within 2 weeks
15. Female, who is pregnant, lactating or planning pregnancy during the study period
16. Has participated in prebiotics or laxative trial within 3 months prior to enrollment or any other clinical trial within 1 month
17. Donated blood within last 3 months
18. Working overnight (e.g. 3rd shift)
19. Excessive coffee and tea consumption (> 4 cups/day)
20. Men and women who do excessive exercise regularly or athlete
21. Men and women whom investigator is uncertain about subject's capability or willingness to comply with protocol requirement

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiome composition as measured by 16S rRNA gene sequencing in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  gut microbiome composition changes

SECONDARY OUTCOMES:
Changes in plasma red raspberry polyphenol metabolites in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  Plasma red raspberry polyphenol metabolites
Changes in insulin sensitivity as measured by the Matsuda composite index of insulin sensitivity (MISI) in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  Plasma Insulin Sensitivity
Changes in plasma glucose response in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  Plasma glucose response
Changes in plasma insulin response in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  plasma insulin response
Changes in urine creatinine concentration in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  urine creatinine concentration
Changes in urine red raspberry polyphenol metabolites in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  urine red raspberry polyphenol metabolites
Changes in breath hydrogen exhalation in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  breath hydrogen exhalation
Changes in Gastrointestinal Health as measured by Gastrointestinal Tract Questionnaire in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  Gastrointestinal Health
Changes in blood pressure in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  blood pressure

OTHER OUTCOMES:
Changes in body weight in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  body weight
Changes in waist circumference in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  waist circumference
Changes in plasma triglycerides in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  plasma triglycerides
Changes in plasma LDL cholesterol in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  plasma LDL cholesterol
Changes in plasma HDL cholesterol in 12-week intervention of active treatment vs Experimental | baseline, 4 weeks, 8 weeks and 12 weeks
  plasma HDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Britt M Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang X, Zhao A, Sandhu AK, Edirisinghe I, Burton-Freeman BM. Red Raspberry and Fructo-Oligosaccharide Supplementation, Metabolic Biomarkers, and the Gut Microbiota in Adults with Prediabetes: A Randomized Crossover Clinical Trial. J Nutr. 2022 Jun 9;152(6):1438-1449. doi: 10.1093/jn/nxac037. PMID 35421233